CLINICAL TRIAL: NCT02411955
Title: A Multiple-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.1% to Tazorac® (Tazarotene Cream 0.1%) and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing Tazarotene Cream 0.1% to Tazorac® and Both to a Placebo Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAZC 1308
Record Dates: First submitted 2015-04-04; First posted 2015-04-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tazarotene Cream 0.1% (Experimental): Tazarotene Cream 0.1% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Tazarotene Cream 0.1%
- Tazorac® (Active Comparator): Tazorac® (tazarotene cream 0.1%) (Allergan LLC)
  Interventions: Drug: Tazorac®
- Placebo (Placebo Comparator): Placebo (Vehicle of the test product) (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tazarotene Cream 0.1% — Tazarotene Cream 0.1% applied to lightly cover the entire face once daily for 84 consecutive days.
  Other Names: Tazarotene
  Arms: Tazarotene Cream 0.1%
Drug: Tazorac® — Tazorac® applied to lightly cover the entire face once daily for 84 consecutive days.
  Other Names: Tazarotene
  Arms: Tazorac®
Drug: Placebo — Placebo (vehicle of the test product) applied to lightly cover the entire face once daily for 84 consecutive days.
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the therapeutic equivalence and safety of Tazarotene Cream 0.1% and Tazorac® (tazarotene cream 0.1%).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the therapeutic equivalence and safety of Tazarotene Cream 0.1% and Tazorac® (tazarotene cream 0.1%) in the treatment of acne vulgaris and to demonstrate the superiority of the test and reference products over the placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects aged 18 years and older must have provided written consent. Subjects aged 12 to 17 years must have provided written assent accompanied by written consent from their legally acceptable representative. All subjects or their legally acceptable representatives must sign Health Insurance Portability and Accountability Act authorization.
* Must have a minimum of ≥ 25 non-inflammatory lesions and ≥ 20 inflammatory lesions and ≤ 2 nodulocystic lesions at baseline on the face.
* Must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Have a history of hypersensitivity or allergy to tazarotene, retinoids and/or any of the study medication ingredients.
* Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1077 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts
Change in non-inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts

SECONDARY OUTCOMES:
Clinical response of success | Week 12
  The proportion of subjects with a clinical response of success at week 12, success defined as an Investigator's Global Assessment score that is at least two grades less than the baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No